CLINICAL TRIAL: NCT02842957
Title: An Intensive Lifestyle Intervention Program in CKD (Move to Health 2)
Acronym: MTHL2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Springfield College (Other)
Collaborators: Relypsa, Inc. (Industry)
Responsible Party: Principal Investigator, Samuel A. Headley, Professor of Exercise Science, Springfield College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Move to Health 2
Record Dates: First submitted 2016-07-18; First posted 2016-07-25 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Kidney Disease
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle intervention (Experimental): Behavioral: The Lifestyle arm is the experimental group that will be exposed to an intensive, individualized approach aimed at assisting these CKD patients to adhere to lifestyle changes that are expected to be beneficial to their health and wellbeing. Patients will receive direction to implement a plant based diet, along with more physical activity in their lives. They will be assisted with the optimal use of their prescribed medications by pharmacy professionals and they will receive behavioral counseling by experts in that area.
  Interventions: Behavioral: Lifestyle Intervention
- Usual Care (No Intervention): The Usual Care arm will continue to receive the current standard of care involving all the services provided at a contemporary nephrology practice in Western Massachusetts

INTERVENTIONS:
Behavioral: Lifestyle Intervention — Patients randomized to the lifestyle group will be given individual counseling regarding the implementation of a plant based diet. They will also be given a home based exercise program to complete. Patients will be assisted with the optimal use of their prescription medications and they will receive specific counseling regarding strategies to help them successfully change their behavior.
  Arms: Lifestyle intervention

SUMMARY:
The primary purpose of the current 6-month study is to determine the effect of an integrated, comprehensive, individualized, intervention program including dietary, exercise, pharmacy, and behavioral counseling on patient performance of the short physical performance battery (SPPB) which gives an indication of an individual's ability to perform activities of daily living dependent upon lower extremity function. Additional objectives include the impact of the intervention on cardiovascular risk factors, and the impact of the intervention on other indices of physical function in stage 3-4 CKD patients. The investigators hypothesize that patients who participate in this integrated, intensive, individualized lifestyle intervention will have higher SPPB scores compared to individuals in the usual care group. The investigators also hypothesize that this approach will lead to higher adherence rates to the lifestyle recommendations and that those who adhere will also show better improvements in the measured variables over time compared to patients who are randomly assigned to the usual care group or who comply poorly with the various study components.

DETAILED DESCRIPTION:
The study will be advertised at Renal and Transplant Associates of New England (RTANE) and interested patients will be screened and cleared by nephrologists from RTANE to make sure that they do not have any contraindications to exercise as described by the American College of Sports Medicine. Those patients who are eligible (stage 3-4, eGFRs 15-59 ml/min/1.73m2) to participate, and who want to be involved , will be asked to read and sign a consent form, which had been reviewed and approved by the Institutional Review Board of Springfield College. This signing will take place at RTANE prior to coming to the College.

Individuals will be randomly assigned to either the lifestyle intervention group or the usual care group. During the course of the study, serum potassium levels will be monitored on a monthly basis in all patients. For individuals randomized to the intervention group, if their levels are greater than 5.2 mEq/L, these patients will be prescribed Veltassa according to the recommended dosing scheme. Individuals randomized to the usual care group will be under the care of their physicians and will receive the current standard of care. They will be able to take Veltassa, if prescribed by their physician, but this will not be required by the study protocol. At baseline, and at month 6, when the blood samples are taken for potassium assessment, some of the sample will also be used for the assessment of other biomarkers that will be tracked in this study (e.g., phosphorus, inflammatory markers, etc) After 6 months of participation in the study, individuals will be retested with the same protocols used at baseline.

Pretest instructions: Following the signing of the consent form, patients will be given instructions as to how to complete a 3-day diet log. Patients will be asked to complete the Exercise Benefits/Barriers Scale (EBBS) and they will be expected to send these completed forms to the faculty at Springfield College prior to arriving at the College for their day-long program.

Program Day: Patients will be expected to come to Springfield College on a Saturday and participate in the program from 8:45 am to approximately 4 PM depending upon their group assignment. Upon arrival at the College, participants will be asked to have all the medications and over-the-counter drugs documented by clinical Pharm D researchers. Any participants who had not previously submitted their dietary information prior to coming will be asked to submit their logs at that time and a member of the research team will take their records and analyze them during the time while they are undergoing the other assessments.

Assessments

During the morning period all patients are assessed for the following variables:

Anthropometrics: Anthropometric measurements including height and weight will be taken. Waist girth will be assessed using a tension tape measure (Gulick) while body composition will be assessed using bioelectric impedance analysis (Tanita, model BC-418).

Cardiovascular assessments: Prior to performing any activity assessment for the day, patients will have their resting blood pressure determined, in their dominant arm, using a calibrated automated sphygmomanometer (Tango, Sun Tech Medical, Morrisville, NC). They will also have pulse wave analysis (PWA) performed on them using a Sphymocor machine (EXCEL). This will give information about their augmentation index (a measure of arterial stiffness), along with a measure of their central blood pressure and pulse pressure.

Functional Movement Screen (FMS): Each participant will be assessed on their ability to perform each of the following movements without restriction: deep squat, active straight leg raise, shoulder mobility, trunk stability push up. A score is assigned based upon how well these movements are performed.

Functional tests: Following the anthropometric assessments, a series of functional tests will be administered. The six minute walk test will be performed with each participant according to American Thoracic Society guidelines. A 20-meter, flat hallway will be used as the course with cones set at each end as a marker. Every 3 feet will be marked along the course. Chairs will be available to the participants at both ends of the course, as well as the middle distance mark. Participants will be instructed to complete the most distance in the time allotted, only walking. At each minute, the participants will be told "You are doing well, you have 5 (4, 3, 2, 1) minutes to go." When 15 seconds are left, the participants will be told to wait for a "Stop" command and instructed to stop wherever they are on the course. The partial lap distance will then be recorded and added to the total lap distance.

The sit-to-stand-to-sit test will also be used for all participants. A sturdy, armless chair with a height of 43.7 cm will be used. Each participant will be instructed to fold their hands over their chest and complete one practice sit-to-stand-to-sit. It will be made clear that no hands are allowed to be used. Then, each participant will be instructed to sit up and down ten times as fast as they can and the time to complete this will be recorded in seconds.

A Short Physical Performance Battery (SPPB) score will be created by summation of the scores for tests of standing balance, gait speed, and rising from a chair 5 times. The SPPB has been shown to have excellent reliability and predictive validity for a number of outcomes including mortality, onset of disability, and institutionalization, and has been used in large, multicenter, randomized controlled trials and observational studies as a primary outcome and for screening purposes.

Grip Strength: Grip strength will be assessed using a Jamar hand held dynamometer. Participants will be asked to sit in a chair while flexing their dominant arm to a 90° angle. The dynamometer will be fitted to each individual's hand and then each participant will be asked to exert maximal effort three times. The highest recorded score (in kg) will be used in statistical analyses.

Strength/Power Assessments: Baseline strength and power will also be assessed with the dominant leg (quadriceps and hamstrings) using isokinetic dynamometry (Biodex). The purpose of the test will be explained to the participants. Each participant will then be strapped into the seat securely using chest straps, a lap strap and leg strap. The straps are to ensure no accessory muscles are used during the test. The participant will then be adjusted into the machine so that the fulcrum of the lateral aspect of the dominant knee is exactly aligned with axis or rotation on the machine. All baseline adjustments will be recorded for each participant at this point. Once the participant is ready to engage, their information regarding ROM and weight of the limb will be adjusted according to computer program procedures. Each participant will be given a trial round of 4 repetitions and will be instructed to push and pull with their leg as hard as they could. Then, 3 rounds of testing will be completed at 5 repetitions for each speed of 90/120/150 degrees per seconds. Each participant will be reminded to breathe, and not hold their breath during the time they are being assessed. Strength and power measurements will then be recorded for each participant.

After these testing sessions are completed, individuals assigned to the usual care group will receive dietary advice and then be allowed to go home while individuals randomized to the intervention groups will be given instructions as to how to prepare a plant-based meal by a professional chef at the College's dining services. Following lunch, each participant will rotate through each of the following stations to receive one-on-one counseling from experts in the specific areas based upon their own specific scores from their earlier assessments. The following section contains information regarding the specific information that will be covered in each of those areas:

Behavioral Methods Instruments: Kidney Disease and Quality of Life (KDQOL) - Short Form (12). The KDQOL-36™ is a short form that includes the SF-12 as generic core supplemented with multi-item scales targeted at particular concerns of individuals with kidney disease (i.e. the burden of kidney disease, symptoms/problems of kidney disease, and effects of kidney disease scales on daily life). The KDQOL-SF is derived from the KDQOL(13), the long-form of the questionnaire, whose use is limited by its length (134 items). The questionnaire is one of the most complete instruments currently available to assess the health related quality of life (HRQOL) of patients because it includes general and specific aspects of health, allowing a more complete evaluation of HRQOL dimensions that are relevant for the patients . The authors of the KDQOL developed a standalone Excel scoring tool which was used to score the instrument.

The Self-Efficacy to Regulate Exercise Habits Questionnaire. Self-efficacy to regulate exercise habits relates to the belief that one can perform exercise activities in the face of impediments (e.g.., fatigue, time constraints, unfavorable environmental conditions, and competing demands). Subjects will rate themselves on scales that range from 0 ("cannot do"); through intermediate degrees of assurance, 50 ("moderately certain can do"); to complete assurance, 100 ("highly certain can do").

The Self-Efficacy to Regulate Eating Habits Questionnaire (Cronbach alpha = 0.93) Subjects will be asked to rate their confidence in being able to "stick to healthy eating habits" when faced with different tempting situations (e.g. when very hungry, when eating out with others, during holiday times, when feeling upset). Subjects rate themselves on scales that range from 0 ("cannot do"); through intermediate degrees of assurance, 50 ("moderately certain can do"); to complete assurance, 100 ("highly certain can do").

Participants in the intervention conditions will be given brief individualized counselling to achieve their lifestyle goals. Participants will meet one-on-one with a behavioral health counselor to develop their personalized self-management program. A program will be formulated for each patient in which manageable goals for lifestyle change are negotiated, and specific individually tailored intervention strategies to increase self-efficacy and decrease barriers to change will be developed. The key features of the intervention will be a) assessment of current physical activity and dietary habits, b) investigating the perceived benefits, barriers and costs of behavior change, c) patient participation in goal setting and selecting personalized strategies to overcome barriers and prevent relapse, and d) establishing follow-up contacts. Regular self-assessment will be used to empower participants to take responsibility for their own decisions and to make informed choices.

Follow-up contact will be made via email by the same counselor who met with the patient at the assessment visit, at one week post-assessment and monthly thereafter. These emails will focus on the extent to which patients have achieved their goals since last contact, and patients will be reinforced or assisted in problem-solving additional strategies as appropriate. Patients will also receive additional written materials tailored to their current concerns (e.g. focusing on lapse and relapse, discussion of time management strategies, and cues to get back into an activity plan after holidays).

Pharmacy Methods:

A clinical PharmD researcher will conduct patient interviews. Preparation for the interviews include contacting the participants requesting that they bring all prescription and over-the-counter medications to the "Move to Health Study." Patients will be specifically informed to bring all prescription (including those only taken as needed), over the counter medications (such as medicine for sleep, allergies, etc.), vitamins, herbals, creams and inhalers used within the past month.

At the beginning of the Move to Health Study, participants will provide their bag of medications to the pharmacist. While the patients are completing the initial phases of the study, the pharmacist will document each medication including dosage, sig, day's supply and last refill date, and will evaluate each medication for nephrotoxic effects, interactions, contraindications and medication appropriateness in CKD. This will be done for each patient without the pharmacist's knowledge of patient randomization group. Any medication that is identified as potentially harmful or nephrotoxic for any patient will be addressed with the lead physician of the study group for further discussion.

Once patients are randomized, those assigned to the intervention groups will meet individually with the pharmacist. Patients in the usual care group are excused without pharmacy associated changes as long as there are no medications identified as potentially harmful or nephrotoxic. A detailed patient medication history will be obtained, including the current dose; schedule and patient reported side effects. Adherence and associated barriers will be assessed using the Morisky 8-point adherence tool (MMSA-8). Patients will also be asked specifically, "Within the past week, how many doses of medication have you missed?" Based upon the information gathered, the pharmacist will make evidence-based interventions. Interventions include providing each patient with a recommended dosing schedule, appropriate timing in relation to food and other medications, and tools to improve adherence. These tools include recommending pill organizers, timers and decreasing medication dosing frequency. Medication schedule will be based on pharmacokinetic and pharmacodynamics considerations as well as therapeutic guideline recommendations. The administration of the drug will comply with the standard operating procedures followed at RTANE (see attached SOP). The medications will be stored at RTANE in a research refrigerator that is maintained at 2-8 °C temperature and when dispensed to subjects they will be told to do the same. This research refrigerator is monitored to make sure that it is keeping the stored medications at the correct temperature. Patients will be educated about medication indication, OTC and herbal medications to eliminate and to avoid (e.g., NSAIDs). Patients will be provided an opportunity to ask medication related questions that will be addressed individually by the pharmacist.

In the intervention group, the pharmacist will follow the following algorithm which is based on the most recent KDIGO guidelines:

1. If the subject is on a RAS blocker, the pharmacist will titrate the dose up to maximal dose in order to achieve a BP <130/80.
2. If the patient has an elevated urinary albumin excretion, the RAS inhibitor dose will also be titrated to the maximal dose.
3. If the potassium is >5.2, Veltassa will be provided and dosed according to the PI Nutrition Methods Participants will be required to keep a 3-day food log prior to the day-long program. The information from the food logs will be analyzed with a Food Processor Diet Analysis Software program (ESHA, Salem, OR) for nutritional content. The ESHA Food Processor Nutrition Analysis software is widely used to assess the nutrient content of food in both research and clinical practice. The software provides analyses for more than 55,000 foods and food items, providing analysis for more than 163 nutritional components.

During the dietary consultation, the diet analysis will be reviewed with the participant, regarding their individual dietary macronutrient and micronutrient content. Specific attention will be paid to the amount and quality of protein, as well as the amount of sodium, phosphorous, and potassium contained in the diet. Recommendations for dietary modifications will be based on a vegan approach. Participants in the intervention group will be encouraged to decrease the amount of animal protein in their diet and choose more plant-based meals. The quality of animal protein will be addressed; with red meat and dairy products most highly discouraged, followed by poultry, and fish. Education will be provided on the significance of reducing sodium, phosphorous, and potassium on kidney health. Strategies to reduce the intake of these micronutrients will be presented, specifically what types of foods to avoid and what types to include more of in the diet. Individual barriers to success in achieving the suggested dietary modifications will be addressed, and strategies to implement the changes will be discussed based on the participant's individual circumstances. Participants will also attend lunch with a cooking education session, in which a professional chef will demonstrate how to prepare a vegan meal. During this session, strategies to enhance the flavor and appeal of plant-based meals will be presented to aid participants in being able to practically include plant-based meals in their daily diet. The treatment group will have an unrestricted potassium diet. Individuals randomized to the control group will be counseled on a standard 1 gram/kg protein diet with 2 gram potassium and sodium restriction. Dietary adherence will be assessed in the control and intervention group using a food frequency questionnaire (FFQ). A standard portion size and six possible frequency of consumption responses, ranging from "never" to "two or more times per day" will be given for each food group based on food and nutrients emphasized or minimized in the prescribed diet (i.e., animal protein, sodium, and potassium).

Physical fitness methods: Based upon the performance of the FMS, individuals will be counseled with regard to the types of exercises they should perform. The prescribed exercises will be demonstrated and taught to the subjects so that when they leave to go home they know how to perform the exercises in correct form. Examples of exercises that could be demonstrated are as follows:

* Wall hip hinge
* Chair squat
* Dumbbell bent over row
* Seated horizontal band row
* Seated vertical band row
* elevated push up and wall push up
* Seated one arm dumbbell press,
* Band curl,
* Band triceps push down

Each participant will be also given a set of stretches to perform and will be taught how to perform these stretches by the research staff members responsible for fitness. Examples of stretches that could be used are as follows:

* Wall calf stretch
* Seated and standing hamstring stretch
* Chair quadriceps stretch
* Wall chest stretch
* Wall latissimus dorsi stretch. Subjects will also be instructed to aim to walk for at least 30 minutes, 5 times per week at a moderate intensity to comply with standard physical activity recommendations of accumulating at least 150 minutes per week of moderate intensity physical activity. They will be instructed to avoid prolonged periods of time engaging in sedentary behavior by aiming to reduce sitting time. Examples of ways to reduce this sedentary behavior will be discussed with each participant and they will be encouraged to implement strategies that could work for them. Some that could be used include standing during commercial breaks while watching television and consciously taking movement breaks during each hour by setting a timer for 15-20 intervals.

As previously stated, participants in the intervention group will be issued with a packet of exercises to do at home. This packet will contain simple step by step instructions and illustrations of how to perform these movements with correct form. Prior to leaving the College for the day, each of these exercises will be demonstrated to each participant and they will be taught how to perform these exercises in correct form. A member of the research group will contact them (either by phone or email) at the beginning of each week during the intervention period to review with them the exercise program for the week to come and to discuss any challenges that they might have encountered in the previous week. The means of communication used will be decided upon depending upon the preference of the participant. During these weekly communications, the member from the research team will review the strategies the participant has been using to reduce sedentary behavior and provide encouragement in these endeavors. Participants will also be required to keep a log of their activities and return this log to the research team when they return for their retest dates. The activity log serves as a motivational tool and as an aid for the research team to supervise (and adapt if necessary) the exercise program. Participants will be encouraged to contact the research coordinator at any time if they have any questions or need clarification while performing their home-based exercise program.

Physical Activity Monitoring: By the end of the testing day, each participant will be given a GT3XPB Actigraph monitor (Actigraph, Pensacola, FL) with instructions to wear the monitor for the following 7 days. They will then be asked to return this monitor to the research coordinator who will download the data for storage and later analysis. This process will be repeated each time participants come to the College for testing. Objective data captured by the ActiGraph system (i.e., mean times spent in sedentary behavior, light, and moderate to vigorous physical activity) will be used to compare physical activity and sedentary behavior in the intervention and control group as a measure of exercise adherence.

Planned Follow up All participants in the Move to Health Study will be expected to return to the College approximately one, three and 6 months to be reassessed with the identical procedures as performed at the initial visit. Standard CKD labs (CBC, electrolytes, BUN, creatinine, PTH. magnesium, uric acid and urinary albumin excretion) will be measured at each assessment.

Data Storage All study data will be collected and managed using Research Electronic Data Capture) REDCap electronic data capture tools. REDCap is a secure (password protected), web-based application designed to support data capture for research studies, providing: 1) an intuitive interface for validated data entry; 2) audit trails for tracking data manipulation and export procedures; 3) automated export procedures for seamless data downloads to common statistical packages; and 4) procedures for importing data from external sources. The computers on which the electronic data will be stored will be password protected and the PI other members of the research team will know the code. Apart from the PI, graduate students who will help with data entry, under the PI's supervision and the statistician, will be the only individuals who will have access to the data. To maintain subject confidentiality, upon entry into the study subjects will be assigned a number and that number will be linked to their data in the spreadsheet of the statistical program. No names will be directly linked to the data entered into the statistical program. Random checks of the accuracy of the data entered into the statistical package will be done by the study coordinator and the statistician.

ELIGIBILITY:
Inclusion Criteria:

* Must be stage 3-4 of CKD (GFR 15-59 ml/min/1.73m2)
* Must be between the ages of 18-75 years old,
* Must be capable of complying with and following the study protocol(diet and exercise)
* Must be capable of independently giving informed consent

Exclusion Criteria:

* if the patient is currently on Veltassa
* if in an exercise program,
* if the patient suffers from severe constipation,
* if they have bowel obstruction
* if they have impaction
* if the patient has post-operative motility disorders (i.e., GI disorders).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-07; Primary Completion 2017-12-02 (Estimated); Study Completion 2017-12-15 (Estimated)

PRIMARY OUTCOMES:
Physical Function Measure | 6 month intervention
  Short Physical Performance Battery

SECONDARY OUTCOMES:
KDQOL-SF | 6 months
  The KDQOL-36™ is a short form that includes the SF-12 as generic core supplemented with multi-item scales targeted at particular concerns of individuals with kidney disease (i.e. the burden of kidney disease, symptoms/problems of kidney disease, and effects of kidney disease scales on daily life).

CONTACTS AND LOCATIONS:
Locations (1):
- Springfield College, Springfield, Massachusetts, United States